CLINICAL TRIAL: NCT05411432
Title: Clinical Study of 68Ga Labeled HER2 Affibody Analogues in Healthy Volunteers and Patients With Breast or Gastric Tumors
Brief Title: Clinical Study of 68Ga Labeled HER2 Affibody Analogues
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20202093-F-1
Record Dates: First submitted 2022-06-05; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: HER2-positive Breast Cancer and Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: 68Ga labeled HER2 Affibody — inject the tracer to subjects and perform PET/CT scans

SUMMARY:
The purpose of this study is to assess the dosimetric properties of the positron emission tomography (PET) imaging probe 68Ga labeled HER2 Affibody analogues and preliminarily evaluate its diagnosis value in patients with breast or gastric tumors.

DETAILED DESCRIPTION:
6 healthy volunteers with whole-body PET/CT scans at 0-1.0, 2.0, 3.0 and 4.0 hours after tracer injection (mean dose, 4.93 ± 0.10 mCi) will be performed. During the imaging period, 1 mL blood samples will be obtained specifically at 1, 3, 5, 10, 30,60, 90, 120, 150, 180 and 240 minutes after the injection, for time-activity curve calculations. The estimated radiation doses will be calculated by using OLINDA/EXM software.

50 patients with breast or gastric tumors will be enrolled for the clinical study, they will be performed with both 68Ga-HER2 Affibody PET/CT and18F-FDG PET/CT scans before surgery. The preoperative images are compared and correlated with the pathologically report. Next, the expression of HER2 will be determined by immunohistochemical staining of the resected brain tumor tissues.

ELIGIBILITY:
Inclusion Criteria:

* patients with breast or gastric cancers: diagnosed by MR and ready for surgery

Exclusion Criteria:

* refuse or cannot endure surgery pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
SUV of organs | 0, 0.5, 1.0, 2.0,3.0 and 4.0 hours after injection
  The standardized uptake values (SUV) in deferent organs

SECONDARY OUTCOMES:
radioactivity of blood sample | 1, 3, 5, 10, 30,60, 90, 120, 150, 180 and 240 minutes
  blood samples are obtained specifically at 1, 3, 5, 10, 30,60, 90, 120, 150, 180 and 240 minutes after the injection, for time-radioactivity curve calculations.

IPD SHARING:
Plan to Share IPD: No